CLINICAL TRIAL: NCT01630356
Title: Monitoring Secondhand Smoke Exposure in Buildings in Armenia: Controlled Trial
Brief Title: Controlled Trial to Reduce Secondhand Smoke Exposure at Homes in Armenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: American University of Armenia (Other)
Responsible Party: Principal Investigator, Frances Stillman, Ed. D, Johns Hopkins Bloomberg School of Public Health, Department of Health, Behavior and Society, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 00002501
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Tobacco Use and Smoking Behavior
Keywords: Secondhand Smoke; Nicotine; Indoor Air Pollution
MeSH Terms: conditions — Tobacco Use; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: in-person counseling; Device: Demonstration of PM2.5 Pollution; Behavioral: Follow-up Counseling Calls; Behavioral: Printed material
- Control group (Active Comparator)
  Interventions: Behavioral: Printed material

INTERVENTIONS:
Behavioral: in-person counseling — The interventionist provided in person counseling on eliminating child exposure to tobacco smoke to at least one daily smoker and a non-smoker mother in the household. The counseling session emphasized the following issues: a) importance of healthy environment at home, b) health dangers of smoking and exposure to secondhand smoke, c) why and how to quit smoking, and d) how to keep home air smoke-free.
  Arms: Intervention group
Device: Demonstration of PM2.5 Pollution — The study team measured the particulate matter (PM2.5) in the air using the TSI AM 510 Aerosol SidePak to compare the quality of indoor air with outdoor air and demonstrate the effect of smoking on indoor air quality in the intervention households. After completing the Side Pack PM2.5 measurement, the interventionist immediately downloaded the data to a laptop to visualize the results through graphical presentation of the PM2.5 fluctuations to family members.
  Arms: Intervention group
Behavioral: Follow-up Counseling Calls — Interventionists made two follow-up counseling calls to the primary contact in the intervention households, usually a non-smoking mother at one and two months after the in-person counseling session. These calls aimed at a) assessing the progress in meeting the goals set earlier, b) counseling on barriers to the change, and c) encouraging study participants to maintain the success or to set new goals. These calls also provided opportunity for the participants to ask questions or clarify issues
  Arms: Intervention group
Behavioral: Printed material — The intervention group families received the tailored and culturally adjusted educational brochure developed by the study team.
  The control group received a brief educational leaflet on the hazards of SHS developed by the US Environmental Protection Agency.

SUMMARY:
This study was designed to test the hypothesis whether a novel intervention that uses motivational interviewing along with immediate feedback and follow-up counseling calls is effective in educating the household members about the health hazards of smoking and secondhand smoke exposure and reducing children exposure to secondhand smoke at households in Armenia.

The study was a randomized control trial with two arms: intervention and control groups.

The sample population for the study included households with a non-smoking mother and at least one child 2 to 6 years of age residing with at least one daily smoker. The study team recruited the households through pediatrician's offices in polyclinics (primary healthcare facilities) utilizing multistage random sampling. Trained interviewers made two baseline (one week apart) and two 4-month follow-up household visits to conduct measurements, interviews and intervention. Measurements included surveys, air nicotine monitoring in homes and hair samples from children to assess changes in nicotine concentration over time.

SHS concentration was estimated by sampling vapor-phase nicotine using a filter badge treated with sodium bisulfate. Airborne nicotine monitors were used in all homes to measure SHS concentration at baseline and 4 month follow-up. At least one monitor was used in each home, preferably in the main room in which the family congregates.

Personal exposure to SHS in 2-6 years old children was assessed using biological samples of hair. A small sample of hair (approximately 30 - 50 strands, 2-3 cm) was cut near the hair root from the back of the scalp where there is the most uniform growth pattern between individuals which minimizes the variability of the results.

The intervention included an in-person counseling session with distribution of a tailored educational brochure and demonstration/feedback measurement of indoor PM2.5 (at second baseline visit); it also included one and two months follow-up counseling calls. The control group received only a brief educational leaflet on the hazards of second-hand smoke exposure.

ELIGIBILITY:
Inclusion Criteria:

* At least one child 2 to 6 years of age
* Non-smoking mother
* At least one daily smoker
* Child's exposed to second smoke of at least 1 cigarette per day

Exclusion Criteria:

* Mother's pregnancy
* Child's hair less than 2 cm in length after stretching out
* Residing out of Yerevan

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
change in child's hair nicotine concentration | baseline and 4-month follow-up
change in air nicotine concentration | baseline and 4-month follow-up

SECONDARY OUTCOMES:
change in the respondents' knowledge on hazards of smoking and secondhand smoke | baseline and 4-month follow-up
change in frequency of smoking in the presence of the child | baseline and 4-month follow-up
change in household smoking restrictions | baseline and 4-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Frances A Stillman, Ed.D, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- College of Health Sciences, American University of Armenia, Yerevan, Armenia

REFERENCES:
- [Background] Wipfli H, Avila-Tang E, Navas-Acien A, Kim S, Onicescu G, Yuan J, Breysse P, Samet JM; Famri Homes Study Investigators. Secondhand smoke exposure among women and children: evidence from 31 countries. Am J Public Health. 2008 Apr;98(4):672-9. doi: 10.2105/AJPH.2007.126631. Epub 2008 Feb 28. PMID 18309121
- [Background] Al-Delaimy WK. Hair as a biomarker for exposure to tobacco smoke. Tob Control. 2002 Sep;11(3):176-82. doi: 10.1136/tc.11.3.176. PMID 12198265
- [Background] Hovell MF, Meltzer SB, Wahlgren DR, Matt GE, Hofstetter CR, Jones JA, Meltzer EO, Bernert JT, Pirkle JL. Asthma management and environmental tobacco smoke exposure reduction in Latino children: a controlled trial. Pediatrics. 2002 Nov;110(5):946-56. doi: 10.1542/peds.110.5.946. PMID 12415035
- [Background] Emmons KM, Hammond SK, Fava JL, Velicer WF, Evans JL, Monroe AD. A randomized trial to reduce passive smoke exposure in low-income households with young children. Pediatrics. 2001 Jul;108(1):18-24. doi: 10.1542/peds.108.1.18. PMID 11433049
- [Background] Gehrman CA, Hovell MF. Protecting children from environmental tobacco smoke (ETS) exposure: a critical review. Nicotine Tob Res. 2003 Jun;5(3):289-301. doi: 10.1080/1462220031000094231. PMID 12791524
- [Derived] Harutyunyan A, Movsisyan N, Petrosyan V, Petrosyan D, Stillman F. Reducing children's exposure to secondhand smoke at home: a randomized trial. Pediatrics. 2013 Dec;132(6):1071-80. doi: 10.1542/peds.2012-2351. Epub 2013 Nov 4. PMID 24190686